CLINICAL TRIAL: NCT06304688
Title: Effects of a Yoga Program Combined With Diet on Cognitive, Nutritional Status, Mental and Functional Abilities in Older Adults.
Brief Title: Yoga and Diet on Cognitive, Nutritional Status, Mental and Functional Abilities in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén_24
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Aging
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group (CG) will not undergo treatment, which will be evaluated in the pre- and post-phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity, and they will be given the guide of recommendations for the promotion of physical activity.
- Experimental Group (Experimental): The experimental group (EG), after an initial evaluation, will be subjected to a physical training program based on the yoga method, for 12 weeks with 2 weekly sessions (Tuesday and Thursday), with a duration of 45 minutes per session. Once the intervention is finished, you will undergo a final evaluation again to see if there is a difference or not with the results obtained at the beginning. In addition to the yoga intervention, the experimental group received a Mediterranean diet protocol.
  Interventions: Other: Yoga and Mediterranean Diet intervention

INTERVENTIONS:
Other: Yoga and Mediterranean Diet intervention — It will last 12 weeks with a frequency of 2 sessions per week and each lasting 50 minutes.
  * Warm-up phase (10 minutes): Conscious and gentle breathing. Gentle movements of the neck, shoulders, arms and legs to increase blood circulation and flexibility.
  * Training phase (30 minutes): Series of gentle postures adapted to the needs of older adults. Includes standing, sitting and lying postures for relaxation and stretching. It will begin with basic postures and breathing techniques and will gradually advance as participants gain confidence.
  * Return to calm (10 minutes): Deep relaxation in a lying position to integrate the benefits of the practice and promote total relaxation of the body and mind.
  The Mediterranean diet consisted of: i) carbohydrates constitute 50% of the daily intake; ii) fats represented 35%; and iii) proteins represented 15%.
  Arms: Experimental Group

SUMMARY:
Yoga has emerged as a powerful therapeutic practice for enhancing physical and mental health across all age groups, including older adults and younger individuals. For seniors, yoga aids in maintaining flexibility, muscle strength, balance, and posture, thereby reducing the risk of falls and injuries. It also alleviates chronic pain, enhances sleep quality, and mitigates stress and anxiety, contributing to improved overall mental and emotional well-being in this demographic. As individuals age, they undergo physical and mental changes that impact their quality of life. Yoga offers tailored benefits for older adults by preserving joint mobility and flexibility, lowering the risk of falls, and easing chronic pain associated with conditions like arthritis and osteoporosis. Moreover, it fosters stress reduction, anxiety relief, and depression mitigation, fostering emotional equilibrium. The practice of yoga from a young age yields numerous advantages for both physical and mental health, including enhanced concentration, attention, and memory-beneficial qualities for university students. Moreover, yoga aids in stress and anxiety reduction, fosters positive body image, and bolsters self-esteem, contributing to vitality and active aging. Yoga is efficacious in enhancing quality of life and facilitating healthy aging by offering adaptable, gentle exercise that caters to individual needs and limitations. Its mindfulness and body awareness aspects foster a stronger mind-body connection, fostering overall well-being and balance. With its adaptability and accessibility, yoga transcends socioeconomic barriers and physical conditions, making it a viable option for people of all backgrounds. In a society marked by rising stress and lifestyle-related ailments, yoga emerges as an invaluable therapeutic avenue for promoting health and well-being. Its holistic approach and adaptability to individual needs make it an appealing option for individuals seeking sustainable improvements in physical and mental health. Thus, the integration and promotion of yoga as a therapeutic modality in health and wellness domains are warranted. Also, Nutrition plays a fundamental role in the health and well-being of individuals at all stages of life, but it is especially crucial in old age due to the physiological and metabolic changes that occur during the aging process. Maintaining a healthy and balanced diet is essential for providing the necessary nutrients for proper body function, strengthening the immune system, and maintaining the health of bone and cardiovascular structures. Specifically, the Mediterranean diet is a traditional dietary pattern based on foods commonly consumed in Mediterranean regions such as Greece, Italy, and Spain. It is characterized by high consumption of fruits, vegetables, legumes, nuts, whole grains, fish, and olive oil, along with moderate intake of dairy and red wine, and limited con-sumption of red meat and processed products. This eating style has been the subject of numerous scientific studies highlighting its multiple health benefits. Apart from the physical health benefits for older adults, the Mediterranean diet has consistently been associated with positive effects such as reduced risk of cardiovascular pathologies, de-creased chronic diseases and pro-inflammatory factors, as well as contributing to the prevention of obesity and cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, participants will be required to:

* Who are over 65 years old.
* Who do not participate in any physical exercise program.
* Have sufficient physical autonomy to participate in the physical activities required by the study and are able to understand the instructions, programs and protocols of this project.

Exclusion Criteria:

* All participants with contraindications for performing the physical tests will be excluded.
* Diseases that limit cognitive performance and physical activity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
TMT (Trail Making Test) | Up to twelve weeks
  It is used to assess executive function. It measures timed motor and visual tasks, and is divided into two tests: Part A (TMTA), which assesses speed and psychomotor attention and requires connecting consecutively numbered circles; and Part B (TMTB), which tests executive function and requires connecting alternating circles of numbers and letters. Longer completion times indicate poor performance.
SFT (Senior Fitness Test) | Up to twelve weeks
  Instrument used to assess functional abilities. It consists of the following tests: muscle strength (upper and lower limbs), aerobic endurance, flexibility (upper and lower limbs) and agility, 6-minute walk test, Sit-to-foot test using a chair (measures flexibility of the lower body, Try to clasp hands behind your back, Try to get up, walk 8 feet and sit back.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess hand grip strength.
Mindful Attention Awareness Scale (MAAS) | Up to twelve weeks
  It evaluates, in a global way, the dispositional capacity of an individual to be attentive and aware of the experience of the present moment in everyday life. The scale is a 15-item univariate self-report with a view of the mindfulness construct centered on the attention / consciousness variable.
Digit symbol substitution test (DSST) | Up to twelve weeks
  Paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located at the top of the page. The subject copies the symbol in spaces below a row of numbers. The number of correct symbols within the time allowed, usually 90 to 120 seconds, constitutes the score.
D2 test | Up to twelve weeks
  The test measures the speed of processing, the following of instructions and the goodness of execution in a task of discrimination of similar visual stimuli and which, therefore, allow the estimation of attention and concentration. The resulting scores are: - TR, total responses: number of elements attempted in the 14 lines. - TA, total correct answers: number of relevant elements correct. - Or, omissions: numbers of relevant elements attempted but not marked. - C, commissions: number of irrelevant elements marked. - TOT, total effectiveness in the test, that is, TR-(O+C). - CON, concentration index or TA-C. - TR+, line with the highest number of elements attempted. - TR-, line with the lowest number of elements attempted. - VAR, variation or difference index (TR+)-(TR-). The D2 is a useful instrument in research showing a high degree of validity and reliability.
Isaac test | Up to twelve weeks
  Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.
Anxiety and Depression | Up to twelve weeks
  Hospital Anxiety and Depression Scale (HADS). This scale consists of 14 items with 4 response alternatives ranging from 0 to 3 for a total of 0 to 21 points. It has 2 subscales and the score is obtained by adding the scores of each item that make it up, the interpretation criteria being the following: Range of normality (0-7), Possible case of anxiety or depression (8-10) and Case of anxiety or depression (11-21).
Sleep quality | Up to twelve weeks
  Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-assessment questions or items and 5 more to be completed by the person with whom the participant shares a bed or room (although the latter is only used to provide clinical information). These items generate a total score and 7 components or domains: sleep quality; sleep latency; sleep duration; sleep efficiency; sleep disorders; use of sleeping medications; daytime dysfunction. The PSQI total score ranges from 0 to 21, with a higher score indicating poorer sleep quality.
Balance | Up to twelve weeks
  The Tinetti scale was used to measure physical variables of balance, gait, and fall risk [38,39]. This scale is divided into two parts, one measuring static and dynamic balance with 9 items and a maximum score of 17 points, and another measuring gait with 7 items, with a highest score of 12 points. The sum of the two parts is used to assess fall risk. A higher score indicates a lower risk of falling, with 29 being the maximum score achievable. Scores between 19 and 24 points indicate a risk of falls, while scores below 19 indicate low risk.
Nutritional status | Up to twelve weeks
  Changes in participants' nutritional status were assessed using the Mini Nutritional As-sessment (MNA), which is a validated tool for detecting and evaluating malnutrition and the risk of malnutrition in older adults (≥65 years). It consists of 18 questions divided into 4 domains: anthropometric assessment (weight, height, BMI, and arm and calf circum-ferences), global assessment (lifestyle, medication, and mobility), dietary assessment (number of meals and food and liquid intake), and subjective perception of health and nutrition. Each item has a numerical value, and the total score has a maximum value of 30. The MNA classifies nutritional status as adequate (score of 24 to 30), at risk of malnutrition (score of 17 to 23.5), and poor (score less than 17).

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No